CLINICAL TRIAL: NCT05740878
Title: Effect of Local Food-Based Oral Nutritional Supplements (ONS) Containing Immunonutrients in the Form of Anthocyanin and Omega-3 on Nutritional Status and Inflammatory Response in Head and Neck Cancer Patients Receiving Radiotherapy
Brief Title: Administration of ONS Based on Purple Sweet Potato in Head and Neck Cancer Patients With Radiotherapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Brawijaya (Other)
Collaborators: Gadjah Mada University (Other)
Responsible Party: Principal Investigator, Fuadiyah Nila Kurniasari, University of Brawijaya, University of Brawijaya
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: UBrawijaya
Record Dates: First submitted 2023-02-06; First posted 2023-02-23 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Oral Nutritional Supplement
Keywords: oral nutritional supplement; immunonutrient; head and neck cancer; radiotherapy; purple sweet potato
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- immunonutrients ONS (Experimental): the intervention group received ONS which contained immunonutrients (omega 3 and anthocyanin)
  Interventions: Dietary Supplement: immunonutrients oral nutritional supplements
- standard ONS (Active Comparator): the control group received standard ONS (isocaloric)
  Interventions: Dietary Supplement: standard oral nutritional supplements

INTERVENTIONS:
Dietary Supplement: immunonutrients oral nutritional supplements — 1 serving of ONS immunonutrients which is 57 grams of ready-to-brew powder yields 200 ml of a liquid formula containing 251 kcal energy (1.26 kcal/ml), 9 grams protein (14%), 94 mg omega-3, and 20 mg anthocyanins.
  Arms: immunonutrients ONS
Dietary Supplement: standard oral nutritional supplements — 1 serving of standard ONS which is 57 grams of ready-to-brew powder yields 200 ml of liquid formula containing 258 kcal energy (1.26 kcal/ml), 5 g (7.5%) protein , 7 g (24%) fat, 43 g (68%) carbohydrate
  Arms: standard ONS

SUMMARY:
The goal of this clinical trial is to compare the effect of local food-based oral nutritional supplements (ONS) containing immunonutrients (omega-3 and anthocyanins) on nutritional status and inflammatory response in head and neck cancer patients receiving radiotherapy. The main questions it aims to answer are:

* Is there any effect of local food-based oral nutritional supplements (ONS) containing immunonutrients (omega-3 and anthocyanins) on the nutritional status?
* Is there any effect of local food-based oral nutritional supplements (ONS) containing immunonutrients (omega-3 and anthocyanins) on inflammatory response?

Participants will participants will receive ONS in powder form ready to brew as much as 2 servings per day for 3 weeks.

Researchers will compare the effect of giving ONS containing immunonutrients compared to standard ONS to see the effect on nutritional status and inflammatory response

DETAILED DESCRIPTION:
The intervention group received ONS which contained immunonutrients with a composition consisting of purple sweet potato flour, egg white flour, whey protein, olive oil, omega 3 powder, sugar, and creamer. While the control group received a placebo in the form of standard ONS (isocaloric) with a composition of powdered skim milk, coconut oil, sugar, maltodextrin, and creamer.

ELIGIBILITY:
Inclusion Criteria:

1. Participant diagnosed with advanced stage head and neck cancer (stages 3 and 4) who received radiotherapy, both as concurrent and adjuvant or chemoradiotherapy
2. Participant aged 18-80 years
3. Participant can consume food, either through a nasogastric tube (NGT) or orally

Exclusion Criteria:

1. Participant has a milk or egg allergy
2. Participant with comorbid renal impairment and/or diabetes mellitus
3. Participant with poor nutritional status with BMI < 17.0 kg/m2

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2022-03-15 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-05-30 (Estimated)

PRIMARY OUTCOMES:
weight change | immediately after the intervention
  The differences in body weight after and before the intervention was given. Weight in kilograms will be measured with digital scales Omron Type HBF 378.
Body mass index (BMI) | immediately after the intervention
  Calculation of nutritional status using the ratio of body weight (kg) to height squared (m2), where body weight is measured using an digital scales Omron Type HBF 378 and height is measured with a stadiometer.
mid-upper arm circumference (MUAC) | immediately after the intervention
  the circumference of the left upper arm, measured at the mid-point between the tip of the shoulder and the tip of the elbow (olecranon process and the acromion). MUAC is measured using a metline in centimeters.
handgrip strength | immediately after the intervention
  a simple and reliable measurement of maximum voluntary muscle strength, that is measured with handgrip dynamometer in kilograms (kg) unit.

CONTACTS AND LOCATIONS:
Overall Officials: Fuadiyah Nila, MPH, Principal Investigator — Gadjah Mada University
Locations (1):
- dr. Sardjito General Hospital, Yogyakarta, DI Yogyakarta, Indonesia

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-02-01): https://cdn.clinicaltrials.gov/large-docs/78/NCT05740878/Prot_SAP_ICF_000.pdf